CLINICAL TRIAL: NCT04834752
Title: Effect of Histamine 2 Receptor Antagonist (H2RA) and Proton Pump Inhibitor (PPI) on the Positivity Rates and Clinical Outcomes of Coronavirus Disease-19 (COVID-19).
Brief Title: Effect of H2 Receptor Antagonist and Proton Pump Inhibitor on the Positivity Rates and Clinical Outcomes of COVID-19
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Soo-Jeong Cho, Clinical associate professor, Seoul National University Hospital
Other Study IDs: 2102-004-1192
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: COVID-19
Keywords: COVID-19; Proton pump inhibitor; H2 receptor antagonist
MeSH Terms: conditions — COVID-19 | interventions — Pantoprazole; Omeprazole; Esomeprazole; Lansoprazole; Dexlansoprazole; Cimetidine; Nizatidine; Ranitidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients tested for COVID-19: Patients who were tested for COVID-19 nasopharyngeal polymerase chain reaction (PCR)
  Interventions: Other: No intervention (Retrospective Cohort Observational)

INTERVENTIONS:
Other: No intervention (Retrospective Cohort Observational) — History of PPI and H2RA prescription of the participants who were tested for COVID-19 will be reviewed.
  Other Names: PPI: Rabeprazole, Pantoprazole, Omeprazole, Esomeprazole, Lansoprazole, Dexlansoprazole; H2RA: Famotidine, Cimetidine, Nizatidine, Ranitidine

SUMMARY:
This retrospective cohort study aims to evaluate the effect of proton pump inhibitor (PPI) or histamine-2 receptor antagonist (H2RA) on the clinical outcomes and positivity rates of Coronavirus Disease-19 (COVID-19).

DETAILED DESCRIPTION:
Previous researches on the association between the use of PPI and H2RA and the treatment and prevention of COVID-19 have reported inconsistent findings. This study aimed to evaluate the effect of H2 receptor antagonists and proton pump inhibitors on the clinical outcomes and positivity rates of COVID-19 using the Korean National Health Insurance (NHI) data. This is a retrospective cohort study using the NHI COVID-19 dataset, which includes health insurance data of individuals who underwent COVID-19 PCR test in South Korea. This study aims to evaluate the effect of the use of PPI and H2RA on the positivity rates and clinical outcomes of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were tested for COVID-19 using real-time reverse transcriptase PCR assay of nasal and pharyngeal swabs

Exclusion Criteria:

* Record of a new prescription of non-steroidal anti-inflammatory drugs (NSAID) within 1 month of the test date
* Patients who died within 48 hours after test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who were tested for COVID-19 using real-time reverse transcriptase PCR assay of nasal and pharyngeal swabs were included. Data were obtained from the Korean national health insurance claims-based database (COVID-19 research dataset). Individuals with a Record of a new prescription of NSAID within 1 month of the test date were excluded because NSAID users for early pneumonia symptoms may initiated for PPIs or H2 blockers.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 test positivity | Through test completion, an average of 1 day
  Test positivity rates for COVID-19 nasopharyngeal polymerase chain reaction (PCR): number of participants diagnosed with COVID-19 compared to the number participants who were tested for COVID-19
Mortality | 60 days
  Mortality of participants who died after diagnosis of COVID-19 (during the hospitalization or after discharge)

SECONDARY OUTCOMES:
Intensive care unit admission rate | 60 days
  Intensive care unit admission rate of patients who were diagnosed with COVID-19
Mechanical ventilator application rate | 60 days
  Mechanical ventilator application rate of patients who were diagnosed with COVID-19
Oxygen apply rate (Nasal prong, Facial Mask, High flow nasal cannula) | 60 days
  Oxygen apply (Nasal prong, Facial Mask, High flow nasal cannula) rates of patients who were diagnosed with COVID-19
Rates of vasopressor and inotrope use | 60 days
  Rates of vasopressor and inotrope use of patients who were diagnosed with COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No